CLINICAL TRIAL: NCT03088930
Title: A Phase II Trial to Evaluate Crizotinib in the Neoadjuvant Setting in Patients With Surgically Resectable, ALK, ROS1, or MET-oncogene Positive Non-small Cell Lung Cancer
Brief Title: Evaluating Crizotinib in the Neoadjuvant Setting in Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-2025.cc
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant treatment with Crizotinib (Experimental): Patients enrolled in this study will be treated with 6 weeks of induction therapy with crizotinib. On the last day of dosing, patients will then undergo surgical resection. 5 years of follow-up will be done via chart review.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Crizotinib is an oral receptor tyrosine kinase inhibitor of ALK, Hepatocyte Growth Factor Receptor (HGFR, c-Met), and ROS1 (c-ros). Crizotinib will be given as a neoadjuvant therapy before surgical resection. The recommended dose of crizotinib is 250mg orally. Participants on this trial will receive this dose, unless dose modification is necessary.
  Other Names: Xalkori

SUMMARY:
This study will evaluate the efficacy of crizotinib as induction therapy in participants with surgically resectable ALK rearrangement, ROS1 rearrangement, or MET exon 14 mutation positive NSCLC.

DETAILED DESCRIPTION:
Participants with stage IA-IIIA, surgically resectable lung adenocarcinoma with an activating alteration in ALK, ROS1 or MET will receive neoadjuvant treatment with crizotinib. This neoadjuvant treatment will last 6 weeks and on the last day of dosing of crizotinib, participants will undergo surgical resection, followed by 5 years of follow-up via chart review.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IA-IIIA NSCLC by 8th edition AJCC staging (that is deemed to be surgically resectable by a board certified thoracic surgeon.
2. Staging by PET-CT scan and MRI brain showing no evidence of metastatic disease (mediastinoscopy is not required unless imaging is indeterminate and is then considered standard of care)
3. Documented evidence of an ALK rearrangement (by FISH, IHC, or NGS), ROS1 rearrangement (by FISH or NGS), or MET oncogene as defined by MET exon 14 skipping (NGS), MET Y1003X mutation or MET gene fusion (NGS) in NSCLC tumor specimen by a CLIA-approved laboratory.
4. Measurable disease defined by RECIST 1.1 criteria.
5. Life expectancy of at least 24 months.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Age ≥ 18 years
8. Have normal QT interval on ECG evaluation QT corrected Fridericia (QTcF) of ≤ 450 ms in males or ≤ 470 ms in females
9. Adequate organ function:

   * Absolute neutrophil count (ANC) ≥1500/µL
   * Platelets ≥75,000/µL
   * Hemoglobin ≥ 10g/dL
   * AST /ALT ≤ 2.5 x upper limit of normal (ULN)
   * Total serum bilirubin ≤ 1.5 x ULN
   * Serum creatinine ≤ 1.5 x UNL
   * Serum amylase/lipase ≤ 1.5 x UNL
10. Negative serum pregnancy test within 7 days of D1 of treatment in women of child bearing potential.
11. If fertile, willing to use highly effective form of contraception (defined as a combination of at least two of the following methods: condom or other barrier methods, oral contraceptives, implantable contraceptives, intrauterine devices) during the dosing period and for at least 4 months after the dosing period.
12. Ability to provide signed informed consent and willing and able to comply with all study requirements.

Exclusion Criteria:

1. Stage IIIB or IV NSCLC.
2. History or the presence of pulmonary interstitial disease, or drug-related pneumonitis.
3. Malabsorption syndrome or other GI illness that could affect oral absorption of the study drug
4. Inability to swallow oral medications
5. Have significant, uncontrolled or active cardiovascular disease, specifically including but restricted to:

   * Myocardial infarction (MI) within 6 months of trial enrollment
   * Unstable angina within 6 months of trial enrollment
   * Congestive heart failure (CHF) with 6 months prior to trial enrollment
   * Any history of ventricular arrhythmia
   * Cerebrovascular accident or transient ischemic attack within 6 months of D1 of treatment
   * Clinically significant atrial arrhythmia or severe baseline bradycardia defined as resting heart rate < 50 beat per minute
   * Uncontrolled hypertension defined as baseline SBP> 160 and DBP > 100 on 3 separate clinic visits or past history of hypertensive urgency, emergency or encephalopathy
6. Have active infection requiring antibiotics
7. Pregnant or lactating female.
8. Prior treatment with an ALK, ROS1 or MET inhibitor
9. Any prior anticancer therapy for this diagnosis
10. Any active cancer diagnosis (basal or squamous cell cancers allowed) within the last 5 years for which the patient is receiving active therapy or which is untreated. Any cancer diagnosis within the last 5 years that is considered "treated" and/ or on surveillance may be included in the trial.
11. Have any condition or illness that, in the opinion of the investigator would compromise patient safety or interfere with evaluation of the study drug (including but not limited to HIV and HCV)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tejas Patil, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant Treatment With Crizotinib
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants eligible for this study will be newly diagnosed with stage IA-IIIA NSCLC and who harbor an activating alteration in ALK, ROS1, or the MET gene
Arm/Group | Neoadjuvant Treatment With Crizotinib
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 62 [55 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With an Objective Tumor Response Rate
Description: Participants' tumor response to treatment will be compared from initial/pretreatment scan to 6 week scan using RECIST 1.1
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Treatment With Crizotinib
Number analyzed (Participants) | 3
participants | 3

2. Secondary Outcome: The Number of Participants With Pathologic Response Rate
Description: Pathologic response rate is defined as < 50% of viable tumor present histologically in the resected tumor specimen.
Time Frame: 37 months
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Treatment With Crizotinib
Number analyzed (Participants) | 3
Participants | 0
Statistical Analysis 1: Comparison: Neoadjuvant Treatment With Crizotinib; Three subjects enrolled. No statistical analysis completed due to low accrual; Test type: Other; Summary statistics = 0; Three subjects enrolled. No statistical analysis completed due to low accrual

3. Secondary Outcome: Number of Participants With an Objective Response Rate
Description: Number of participants with response rate per RECIST 1.1
Time Frame: 6 weeks post treatment
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Treatment With Crizotinib
Number analyzed (Participants) | 3
participants | 0

4. Secondary Outcome: The Number of Participants With Disease-free Survival (DFS)
Description: DFS is defined as the time from treatment to the first of either disease recurrence or death from any cause.
Time Frame: 37 months
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Treatment With Crizotinib
Number analyzed (Participants) | 3
Participants | 0

5. Secondary Outcome: Overall Survival (OS) Measured in Months
Description: OS is defined as the time from study enrollment to death from any cause.
Time Frame: 37 months
Measure: Median (Full Range); unit: months
Arm/Group | Neoadjuvant Treatment With Crizotinib
Number analyzed (Participants) | 3
months | 37 [0 to 37]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Neoadjuvant Treatment With Crizotinib
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Treatment With Crizotinib (N=3)
Nausea (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Insomnia (General disorders) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1)
creatinine increased (Blood and lymphatic system disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
blurred vision (Eye disorders) | 2 (2)
headache (General disorders) | 1 (1)
epigastric discomfort (Gastrointestinal disorders) | 1 (1)
bradycardia (Cardiac disorders) | 1 (1)
ALT increased (Blood and lymphatic system disorders) | 1 (2)
dysgeusia (Gastrointestinal disorders) | 1 (1)
dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
fatigue (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT03088930/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT03088930/ICF_002.pdf